CLINICAL TRIAL: NCT00467168
Title: Effects of Fatty Acid Composition Ratios of Oral Fatty Loads on the Dynamic Metabolism of Postprandial Lipid and Triglyceride-Rich Lipoproteins in Chinese NIDDM Out-Patients
Brief Title: Optimal Dietary Fat Pattern to Prevent Cardiovascular Disease Among Type 2 Diabetes
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Sun Yat-sen University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 522301118
Record Dates: First submitted 2007-04-26; First posted 2007-04-27 (Estimated); Last update posted 2007-04-27 (Estimated); Status verified 2007-04

CONDITIONS: Type 2 Diabetes Mellitus
Keywords: dietary fatty acid composition; postprandial; triglyceride-rich lipoprotein; type 2 diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Diet

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Behavioral: Diet

SUMMARY:
Cardiovascular complications are the leading cause of death among type 2 diabetic patients. Postprandial triglyceride-rich lipoproteins (ppTRLs) are atherogenic. Dietary fatty acid quality, that is, dietary fatty acid composition is related to atherogenesis. However, to date, the overall influence of dietary fatty acid compositions on lipids in different subfractions of ppTRLs still remains unknown among Chinese diabetic patients. This paucity of evidence may limit the establishment of optimal recommendation of dietary fatty acid composition for type 2 diabetes. We have 2 hypotheses:

1. Different dietary fatty acid compositions lead to differential overall responses of lipids in four subfractions of ppTRLs over postprandial 6 h.
2. One dietary fatty acid composition will be identified as anti-atherogenesis for future study as it can improve atherogenic ppTRLs.

DETAILED DESCRIPTION:
Atherosclerosis is the leading cause of death and disability among patients with type 2 diabetes mellitus. These patients characteristically have hypertriglyceridemia, high VLDL and low HDL-cholesterol in the fasting status. During day-time hours, most individuals are in a postprandial state and the composition of postprandial lipoproteins may play a more important role on metabolic outcome than fasting levels. Postprandial triglyceride-rich lipoproteins (ppTRLs) are atherogenic, and longer residence time and higher concentrations of chylomicron and VLDL remnants in the circulation are significant predictors of coronary heart disease (CHD). Abnormal postprandial lipemia is highly prevalent in diabetic patients, even in individuals with a normal fasting triglyceride concentration. It has been suggested that diabetes mellitus is associated with decreased catabolism of chylomicron remnants, prolonged residence of chylomicron and VLDL remnants in the circulation. Therefore, a diet with favorable effects on ppTRLs should be useful to prevent atherosclerosis among type 2 diabetes patients.

It is well known that dietary saturated fatty acids (SFA) increase the risk for CHD while monounsaturated fatty acids (MUFA) and polyunsaturated fatty acids (PUFA) decrease the risk for CHD via the modification of fasting lipids. Since all dietary sources of fat are composed of a combination of SFA, MUFA nad PUFA, it is best to characterize dietary fats as ratio of SFA:MUFA:PUFA. In fact, the SFA:MUFA:PUFA ratio in any given region or population is relatively homogeneous due to common food sources, food accessibility, food preparation and processing, dietary culture and tradition. For example, dietary fatty acid compositions (SFA:MUFA:PUFA) obtained directly or derived from existing national/regional reports are: 1:1.7:0.4 in Greece,1:1.0:0.5 in USA, and 1:1.5:1 in the mainland of China. Our research showed that the composition was 1:1.7:1.2 among type 2 diabetic patients in Guangzhou, a city in Southern China(10). To date, the overall influence of dietary fatty acid compositions on lipids in different subfractions of ppTRLs still remains unclear. This paucity of evidence may limit the establishment of optimal recommendation of dietary fatty acid composition for type 2 diabetes.

We designed three fat loads with specific fatty acid composition based on our previous study and current nutrition knowledge, and aimed at elucidating the influence of these dietary fatty acid compositions on the overall response of lipids in ppTRLs over postprandial 6 h.Based on the result, we will identify on one dietary fatty acid compositions, which can improve atherogenic ppTRLs and thus may be recommended for diabetic patients, for future large-scale research.

ELIGIBILITY:
Inclusion Criteria:

* Type 2 diabetes;
* Types and doses of antidiabetic agents had been unchanged for four weeks before the postprandial study;
* Nonsmokers;
* No prior cardiovascular disease, hepatic and renal diseases, or other diseases influencing fat absorption;
* No previous history of gastro-enteral surgery;
* Dietary fat provided energy less than 35% in last two weeks;
* No use of medications or vitamins known to affect plasma lipids;
* Ability to hold hypoglycemic drugs on the day of the study until postprandial tests are completed;
* Ability to provide verbal informed consent to participate.

Exclusion Criteria:

* Females with menstrual cycles

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 30
Dates: Start 1998-01; Study Completion 1998-05 (Actual)

PRIMARY OUTCOMES:
Lipids including triglyceride and cholesterol in four subfractions of ppTRLs.

SECONDARY OUTCOMES:
Apolipoproteins including apoB100 and apoA1 in the postprandial plasma
Lipoproteins including high- and low-density lipoproteins in the postprandial plasma
Lipids lipoproteins in the postprandial plasma

CONTACTS AND LOCATIONS:
Overall Officials: Jun Dai, MD, Principal Investigator — Department of Clinical Nutrition, School of Public Health, Sun Yat-sen University, Guangzhou, China
Locations (2):
- China (2):
  - Department of Clinical Nutrition, School of Public Health, Sun Yat-sen University, Guangzhou, Guangdong
  - Department of Endocrinology, The First Hospital, Sun Yat-sen University, Guangzhou, Guangdong

REFERENCES:
- [Background] Groot PH, van Stiphout WA, Krauss XH, Jansen H, van Tol A, van Ramshorst E, Chin-On S, Hofman A, Cresswell SR, Havekes L. Postprandial lipoprotein metabolism in normolipidemic men with and without coronary artery disease. Arterioscler Thromb. 1991 May-Jun;11(3):653-62. doi: 10.1161/01.atv.11.3.653. PMID 2029503
- [Background] Mero N, Syvanne M, Eliasson B, Smith U, Taskinen MR. Postprandial elevation of ApoB-48-containing triglyceride-rich particles and retinyl esters in normolipemic males who smoke. Arterioscler Thromb Vasc Biol. 1997 Oct;17(10):2096-102. doi: 10.1161/01.atv.17.10.2096. PMID 9351377
- [Background] Chen J, Gao J. The Chinese total diet study in 1990. Part II. Nutrients. J AOAC Int. 1993 Nov-Dec;76(6):1206-13. PMID 8286957
- [Background] Karpe F, Steiner G, Uffelman K, Olivecrona T, Hamsten A. Postprandial lipoproteins and progression of coronary atherosclerosis. Atherosclerosis. 1994 Mar;106(1):83-97. doi: 10.1016/0021-9150(94)90085-x. PMID 8018110
- [Background] Karpe F, Steiner G, Olivecrona T, Carlson LA, Hamsten A. Metabolism of triglyceride-rich lipoproteins during alimentary lipemia. J Clin Invest. 1993 Mar;91(3):748-58. doi: 10.1172/JCI116293. PMID 8450056
- [Background] Karpe F, Tornvall P, Olivecrona T, Steiner G, Carlson LA, Hamsten A. Composition of human low density lipoprotein: effects of postprandial triglyceride-rich lipoproteins, lipoprotein lipase, hepatic lipase and cholesteryl ester transfer protein. Atherosclerosis. 1993 Jan 4;98(1):33-49. doi: 10.1016/0021-9150(93)90221-f. PMID 8457249
- [Background] Higashi K, Ishikawa T, Shige H, Tomiyasu K, Yoshida H, Ito T, Nakajima K, Yonemura A, Sawada S, Nakamura H. Olive oil increases the magnitude of postprandial chylomicron remnants compared to milk fat and safflower oil. J Am Coll Nutr. 1997 Oct;16(5):429-34. doi: 10.1080/07315724.1997.10718709. PMID 9322191
- [Background] Heyden S. Polyunsaturated and monounsaturated fatty acids in the diet to prevent coronary heart disease via cholesterol reduction. Ann Nutr Metab. 1994;38(3):117-22. doi: 10.1159/000177801. PMID 7979164
- [Background] Brouwer CB, de Bruin TW, Jansen H, Erkelens DW. Different clearance of intravenously administered olive oil and soybean-oil emulsions: role of hepatic lipase. Am J Clin Nutr. 1993 Apr;57(4):533-9. doi: 10.1093/ajcn/57.4.533. PMID 8460608
- [Background] de Bruin TW, Brouwer CB, van Linde-Sibenius Trip M, Jansen H, Erkelens DW. Different postprandial metabolism of olive oil and soybean oil: a possible mechanism of the high-density lipoprotein conserving effect of olive oil. Am J Clin Nutr. 1993 Oct;58(4):477-83. doi: 10.1093/ajcn/58.4.477. PMID 8379502
- [Background] Levy E, Roy CC, Goldstein R, Bar-On H, Ziv E. Metabolic fate of chylomicrons obtained from rats maintained on diets varying in fatty acid composition. J Am Coll Nutr. 1991 Feb;10(1):69-78. doi: 10.1080/07315724.1991.10718129. PMID 2010582
- [Background] Bjorkegren J, Packard CJ, Hamsten A, Bedford D, Caslake M, Foster L, Shepherd J, Stewart P, Karpe F. Accumulation of large very low density lipoprotein in plasma during intravenous infusion of a chylomicron-like triglyceride emulsion reflects competition for a common lipolytic pathway. J Lipid Res. 1996 Jan;37(1):76-86. PMID 8820104
- [Background] Tatami R, Mabuchi H, Ueda K, Ueda R, Haba T, Kametani T, Ito S, Koizumi J, Ohta M, Miyamoto S, Nakayama A, Kanaya H, Oiwake H, Genda A, Takeda R. Intermediate-density lipoprotein and cholesterol-rich very low density lipoprotein in angiographically determined coronary artery disease. Circulation. 1981 Dec;64(6):1174-84. doi: 10.1161/01.cir.64.6.1174. PMID 7296792
- [Background] Tornvall P, Hamsten A, Carlson LA. Abnormalities of composition and of in vitro lipolysis products of human small very low density lipoproteins in hypertriglyceridemia. Atherosclerosis. 1990 May;82(1-2):125-35. doi: 10.1016/0021-9150(90)90151-8. PMID 2360914
- [Background] Reardon MF, Nestel PJ, Craig IH, Harper RW. Lipoprotein predictors of the severity of coronary artery disease in men and women. Circulation. 1985 May;71(5):881-8. doi: 10.1161/01.cir.71.5.881. PMID 3986978
- [Background] Bjorkegren J, Hamsten A, Milne RW, Karpe F. Alterations of VLDL composition during alimentary lipemia. J Lipid Res. 1997 Feb;38(2):301-14. PMID 9162750
- [Background] Puppione DL, Kunitake ST, Hamilton RL, Phillips ML, Schumaker VN, Davis LD. Characterization of unusual intermediate density lipoproteins. J Lipid Res. 1982 Feb;23(2):283-90. PMID 7077142
- [Background] Feldman EB, Russell BS, Chen R, Johnson J, Forte T, Clark SB. Dietary saturated fatty acid content affects lymph lipoproteins: studies in the rat. J Lipid Res. 1983 Aug;24(8):967-76. PMID 6631238
- [Result] Dai J, Su Y, Yan F, Liu S, Xu L, Li J. The pattern of diet and dietary fatty acid in type 2 diabetic out-patients investigated with an accurate food frequency method. J Chinese Public Health. 2000;16(1):43-4.
- [Result] Dai J, Su Y, Ling W, Liang Y, Zhong C, Ou X. Study of fatty acids composition ratio of oral fat loads used in postprandial lipids and lipoproteins metabolism. Chinese J Arteriosclerosis. 2000;8(3):8-13.
- [Derived] Dai J, Su YX, Bartell S, Le NA, Ling WH, Liang YQ, Gao L, Wu HY, Veledar E, Vaccarino V. Beneficial effects of designed dietary fatty acid compositions on lipids in triacylglycerol-rich lipoproteins among Chinese patients with type 2 diabetes mellitus. Metabolism. 2009 Apr;58(4):510-8. doi: 10.1016/j.metabol.2008.11.010. PMID 19303972